CLINICAL TRIAL: NCT06967038
Title: Phase Ⅰ-Ⅱa Clinical Study of Chimeric Antigen Receptor Natural Killer Cell Therapy for High-risk Lymphoma Patients With Primary Sjogren's Syndrome
Brief Title: Chimeric Antigen Receptor Natural Killer Cell Therapy for High-risk Lymphoma Patients With Primary Sjogren's Syndrome
Acronym: CAR-NK
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bangdong Gong (Other)
Responsible Party: Sponsor-Investigator, Bangdong Gong, associate chief physician, Shanghai Tongji Hospital, Tongji University School of Medicine
Organization: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tongji Hospital, Shanghai
Record Dates: First submitted 2025-04-22; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Primary Sjogren's Syndrome; Lymphoma
Keywords: primary Sjogren's syndrome; lymphoma; CAR-NK; Dose limiting toxicity
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-NK (Experimental): CAR-NK cell therapy
  Interventions: Biological: CAR-NK cell

INTERVENTIONS:
Biological: CAR-NK cell — Chimeric Antigen Receptor Natural Killer Cell

SUMMARY:
This study is a phase I-II clinical trial of CAR-NK cell therapy for high-risk lymphoma patients with primary Sjogren's syndrome (pSS). The aim is to determine the optimal dose of CAR-NK cells and evaluate the safety and efficacy of increasing doses of iC9/CAR19/IL15 CB-NK cell therapy. Use i3+3 based design to increase dosage. Dose limiting toxicity (DLT) is defined as the occurrence of CRS within 2 weeks after cell infusion, requiring transfer to the intensive care unit, or grade III-IV acute graft-versus-host disease within 40 days after infusion, or grade 3-5 allergic reactions related to CAR-NK cell infusion. For the purpose of i3+3 design, efficacy is defined as a reduction in the high-risk of lymphoma in pSS patients and at least partial relief of dry mouth and eye symptoms on the 30th day after CAR-NK cell infusion.

DETAILED DESCRIPTION:
The dose escalation method adopts the i3+3 design, and CAR-NK cells are tentatively given three doses based on literature: 5 × 10^6/kg body weight, 1 × 10^7/kg body weight, and 5 × 10^7/kg body weight. Plan to enroll 6-12 subjects. If it is necessary to downregulate the dose due to the safety implications of the initial dose of CAR-NK cells, the researchers will together discuss the level of downregulation or administration method. If the current recommended maximum dose level is not confirmed as a possible recommended therapeutic dose, researchers can decide whether to increase it to a higher dose to determine the possible therapeutic dose. During the experiment, dosage adjustments can be made based on the safety and tolerability data of the subjects. Dose limiting toxicity (DLT) is defined as one or more adverse events related to CAR-NK cell therapy occurring in a subject within 45 days after the first infusion of CAR-NK cells. (1) Inflammatory cytokine release syndrome of grade ≥ 3 within 2 weeks.

(2) Allergic reactions of grade 3 or higher within 2 weeks. (3) Organ damage of grade ≥ 3 within 2 weeks (nerve, cardiovascular, lung, genitourinary, gastrointestinal, liver, skin, etc.). (4) Grade ≥ 3 graft-versus-host disease within 45 days. (5) Deaths related to treatment within 45 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age range of 18-70 years old, gender not limited;
2. Diagnosed with primary Sjogren's syndrome, meeting the 2016 ACR/EULAR classification criteria;
3. Persistent enlargement of salivary glands, lymph nodes, liver, or spleen (imaging/or pathology), and at least 2 of the following 4 conditions are met: ① Cryoglobulinemia; ② Low C4; ③ Decreased white blood cells; ④ Positive for anti SSA or anti SSB;
4. Liver and kidney function, defined as S serum GPT<3 times the upper limit of normal; Serum bilirubin and alkaline phosphatase are less than twice the upper limit of normal, and serum creatinine is ≤ 2mg/dl;
5. Normal cognitive function and voluntarily participate in this clinical trial. Signing a written informed consent form. Can follow and complete all trial procedures.

Exclusion Criteria:

1. Pregnant and lactating women;
2. Patients with hepatitis B, hepatitis C, HIV and other virus infections;
3. Highly allergic constitution or history of severe allergies;
4. Patients with a history of other autoimmune diseases;
5. Patients with severe heart failure, respiratory failure, liver dysfunction, kidney failure, persistent bleeding, malignant tumors, and diabetes insipidus;
6. There are other situations where the researcher deems it inappropriate to participate in this clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence of Dose limiting toxicity (DLT) | 45 days
  The dose escalation method adopts the i3+3 design, and CAR-NK cells are tentatively given three doses based on literature: 5×10^6/kg body weight, 1×10^7/kg body weight, and 5×10^7/kg body weight. Plan to enroll 6-12 subjects. Researchers can together decide whether to increase it to a higher dose to determine the possible therapeutic dose. During the experiment, dosage adjustments can be made based on the safety and tolerability data of the subjects, including limiting toxicity type, incidence, and severity of dose limiting toxicity (DLT).
Safety: Incidence and severity of adverse events (AEs) | 45 days
  One or more adverse events are related to CAR-NK cell therapy occurring in a subject within 45 days after the first infusion of CAR-NK cells. (1) Inflammatory cytokine release syndrome of grade ≥ 3 within 2 weeks. (2) Allergic reactions of grade 3 or higher within 2 weeks. (3) Organ damage of grade≥3 within 2 weeks (nerve, cardiovascular, lung, genitourinary, gastrointestinal, liver, skin, etc.). (4) Grade≥3 graft-versus-host disease within 45 days. (5) Deaths related to treatment within 45 days.

SECONDARY OUTCOMES:
cell treatment efficacy | one year
  A change in the high-risk of lymphoma in pSS patients. Physical examination or B-ultrasound or CT scan indicates change in salivary gland, lymph node, liver, and spleen enlargement.
cell treatment efficacy | one year
  At least partial relief of dry mouth and eye symptoms. Two out of three (dryness, pain, and fatigue) visual analog scales (from 0 [best] to 10 [worst]) showed a decrease of 30% or more in scores.
cell treatment efficacy | one year
  (1) Improved saliva flow rate. The normal range for static saliva flow rate is 0.3-0.4 milliliters per minute, while the normal range for stimulated saliva flow rate (such as after chewing stimulation) is 1.5-2.0 milliliters per 5 minutes. (2) Improved emission computer tomography of salivary gland, including bilateral parotid and submandibular gland uptake and excretion function (relative percentage). (3) Improved schirmer experiment. Normally greater than 5 millimeters per minute. (4) Improved corneal fluorescence staining. Abnormal manifestations include punctate coloring, patchy or linear coloring, or diffuse coloring.
cell treatment efficacy | one year
  Improvement of Disease Activity Scale. Scoring criteria is EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI). Based on the degree and severity of the lesion, the total score is 51 points, with higher scores indicating more active disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality, China